CLINICAL TRIAL: NCT05521087
Title: A Phase I/Ib Study of JNJ-75276617 in Combination With Conventional Chemotherapy for Pediatric and Young Adult Participants With Relapsed/Refractory Acute Leukemias Harboring KMT2A, NPM1, or Nucleoporin Gene Alterations
Brief Title: A Study of JNJ-75276617 in Combination With Conventional Chemotherapy for Pediatric and Young Adult Participants With Relapsed/Refractory Acute Leukemias
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109192; 75276617ALE1003 (Other: Janssen Research & Development, LLC); 2022-000380-46 (EudraCT Number)
Record Dates: First submitted 2022-08-29; First posted 2022-08-30 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Acute Leukemias; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Acute Leukemia of Ambiguous Lineage
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute | interventions — fludarabine; Cytarabine; Dexamethasone; Vincristine; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: <2 Years Old (Experimental): Participants aged less than (<) 2 years old in dose escalation portion of the study will receive JNJ-75276617 orally on a 28-day cycle. Starting dose of JNJ-75276617 is based on the adult dose from the ongoing study NCT04811560 with additional dose reductions based on age. Further dose levels will be escalated based on the dose limiting toxicities (DLT) evaluation by study evaluation team (SET) until the recommended Phase 2 Doses (RP2Ds) has been identified. Participants in dose expansion portion of the study will receive JNJ-75276617 orally at one of the RP2D(s) determined in dose escalation portion of the study, in 3 cohorts divided on the basis of disease diagnosis. Participants with acute myeloid leukemia (AML) and B-cell acute lymphoblastic leukemia (ALL) will receive conventional chemotherapy backbone regimen (dexamethasone, vincristine, pegaspargase, fludarabine, cytarabine and intrathecal chemotherapy) in combination with JNJ-75276617.
  Interventions: Drug: JNJ-75276617; Drug: Fludarabine; Drug: Cytarabine; Drug: Intrathecal Chemotherapy; Drug: Dexamethasone; Drug: Vincristine; Drug: Pegaspargase
- Arm B: >=2 Years Old (Experimental): Participants aged greater than or equal to (>=) 2 years old in dose escalation portion of the study will receive JNJ-75276617 orally on a 28-day cycle. Starting dose of JNJ-75276617 is based on the adult dose from the ongoing study NCT04811560 with additional dose reductions based on age. Further dose levels will be escalated based on the DLT evaluation by SET until the RP2Ds has been identified. Participants in dose expansion portion of the study will receive JNJ-75276617 orally at one of the RP2D(s) determined in dose escalation portion, in 3 cohorts divided on the basis of disease diagnosis. Participants with AML and B-cell ALL will receive conventional chemotherapy backbone regimen (dexamethasone, vincristine, pegaspargase, fludarabine, cytarabine and intrathecal chemotherapy) in combination with JNJ-75276617.
  Interventions: Drug: JNJ-75276617; Drug: Fludarabine; Drug: Cytarabine; Drug: Intrathecal Chemotherapy; Drug: Dexamethasone; Drug: Vincristine; Drug: Pegaspargase

INTERVENTIONS:
Drug: JNJ-75276617 — JNJ-75276617 will be administered orally.
Drug: Fludarabine — Fludarabine chemotherapy will be administered as intravenous (IV) infusion for participants with AML.
Drug: Cytarabine — Cytarabine chemotherapy will be administered as IV infusion for participants with AML.
Drug: Intrathecal Chemotherapy — Intrathecal chemotherapy will be administered as IV infusion for participants with AML or B-cell ALL.
Drug: Dexamethasone — Dexamethasone chemotherapy will be administered as IV infusion for participants with B-cell ALL.
Drug: Vincristine — Vincristine chemotherapy will be administered as IV infusion for participants with B-cell ALL.
Drug: Pegaspargase — Pegaspargase chemotherapy will be administered as IV infusion for participants with B-cell ALL.

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose(s) (RP2Ds) of JNJ-75276617 in combination with a conventional chemotherapy backbone in pediatric and young adult participants with relapsed/refractory acute leukemia harboring histone-lysine N-methyltransferase 2A1 ([KMT2A1], nucleophosmin 1 gene (NPM1), or nucleoporin alterations in Part 1 (Dose Escalation) and to further evaluate safety at the RP2D(s) of JNJ-75276617 in combination with chemotherapy in pediatric and young adult participants with relapsed/refractory acute leukemia harboring KMT2A1, NPM1, or nucleoporin alterations and safety at the RP2D(s) of JNJ-75276617 as monotherapy in a select low burden of disease cohort in Part 2 (Dose Expansion).

ELIGIBILITY:
Inclusion Criteria:

* Acute leukemia harboring histone-lysine N-methyltransferase 2A (KMT2A) or nucleophosmin 1 gene (NPM1) or nucleoporin (NUP98 or NUP214) alterations
* Performance status greater than or equal to (>=) 50 by lansky scale (for participants less than [<] 16 years of age) or >=50 percent (%) karnofsky scale (for participants >=16 years of age)
* Estimated or measured glomerular filtration rate >= 60 milliliter per minute per 1.73 meter square (mL/min/1.73m^2) based on the bed side schwartz formula

Exclusion Criteria:

* Received an allogeneic hematopoietic transplant within 60 days of screening
* Active acute graft-versus-host disease of any grade or chronic graft-versus-host which is not well-controlled
* Received immunosuppressive therapy post hematopoietic transplant within 30 days of enrollment
* Diagnosis of Down syndrome associated leukemia, acute promyelocytic leukemia, juvenile myelomonocytic leukemia
* Diagnosis of fanconi anemia, kostmann syndrome, shwachman diamond syndrome, or any other known bone marrow failure syndrome
* Prior exposure to menin-KMT2A inhibitors
* Prior cancer immunotherapy (ie [that is], Chimeric Antigen Receptor-T Cell Therapy [CAR-T], inotuzumab, gemtuzumab ozogamicin) within 4 weeks prior to enrollment or blinatumomab within 2 weeks prior to enrollment. Additional prior cancer therapies must not be given within 4 weeks prior to enrollment or 5 half-lives of the agent (whichever is shorter)

Ages: 30 Days to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-26 (Estimated); Primary Completion 2026-09-11 (Estimated); Study Completion 2030-01-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 3 years 5 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity | Up to 3 years 5 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Number of Participants with Dose-Limiting Toxicity (DLT) | Cycle 1 (28 days)
  Percentage of participants with DLT will be assessed. The DLTs are specific adverse events related to JNJ-75276617 and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.

SECONDARY OUTCOMES:
Plasma Concentration of JNJ-75276617 | Up to 3 years 5 months
  Plasma concentration of JNJ-75276617 will be reported.
Number of Participants with Depletion of Leukemic Blasts | Up to 3 years 5 months
  Number of participants with depletion of leukemic blasts will be reported.
Number of Participants with Differentiation of Leukemic Blasts | Up to 3 years 5 months
  Number of participants with differentiation of leukemic blasts will be reported.
Changes in Expression of Menin-histone-lysine N-methyltransferase 2A (KMT2A) Target Genes or Genes Associated With Differentiation | Up to 3 years 5 months
  Changes in expression of menin-histone-lysine N-methyltransferase 2A (KMT2A) target genes or genes associated with differentiation will be reported.
Overall Response Rate (ORR) per Response Criteria in Acute Myeloid Leukemia (AML) | Up to 3 years 5 months
  ORR is defined as the percentage of participants who achieve complete response (CR), CR with incomplete hematologic recovery (CRi) or CR with partial hematologic recovery (CRh) per the Response Criteria in AML.
Overall Response Rate (ORR) per the Response Criteria in B-cell Acute Lymphoblastic Leukemia (ALL) | Up to 3 years 5 months
  ORR in participants with B-cell ALL is defined as the percentage of participants who achieve CR or CRi per the response criteria in B-cell ALL.
Time to Response (TTR) | Up to 3 years 5 months
  TTR is defined for the responders as the time from the date of the first dose of JNJ-75276617 to the date of the first documented response.
Duration of Response (DOR) | Up to 3 years 5 months
  DOR will be calculated among responders from the date of initial documentation of a response to the date of first documented evidence of relapse, as defined in the disease-specific response criteria, or death due to any cause, whichever occurs first.
Percentage of Participants With Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) | Up to 3 years 5 months
  Percentage of participants who receive an allogeneic HSCT after treatment will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency